CLINICAL TRIAL: NCT03455777
Title: A Phase 2 Open-Label Study to Assess the Pharmacodynamics, Pharmacokinetics, Safety and Tolerability of ISIS 703802 (AKCEA-ANGPTL3-LRx) Administered Subcutaneously to Patients With Homozygous Familial Hypercholesterolemia (HoFH)
Brief Title: Study of AKCEA-ANGPTL3-LRX (ISIS 703802) in Patients With Homozygous Familial Hypercholesterolemia (HoFH)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn due to lack of available patients meeting entry criteria
Sponsor: Akcea Therapeutics (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 703802-CS4
Record Dates: First submitted 2018-02-22; First posted 2018-03-07 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AKCEA-ANGPTL3-LRX Dose 1 (Experimental)
  Interventions: Drug: AKCEA-ANGPTL3-LRX

INTERVENTIONS:
Drug: AKCEA-ANGPTL3-LRX — Single open-label cohort
  Other Names: ISIS 703802

SUMMARY:
This is a single center, open-label study to evaluate the efficacy of AKCEA-ANGPTL3- LRX for reduction of low density lipoprotein cholesterol (LDL-C) levels in patients with Homozygous Familial Hypercholesterolemia (HoFH).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≤ 35 kg/m2,
* Genetic confirmation of two mutant alleles at the LDLR, APOB, PCSK9, or LDLRAP1 gene locus OR an untreated LDL-C > 500 mg/dL (13 mmol/L) or treated LDL-C ≥ 300 mg/dL (2.59 mmol/L) together with either cutaneous or tendon xanthoma before age 10 years OR familial medical history of genetically confirmed heterozygous FH in both parents OR untreated elevated LDL-C and TC > 250 mg/dL consistent with the disease,
* Patients must be on stable LDL-C lowering agents or on regular apheresis

Exclusion Criteria:

* Myocardial infarction, percutaneous transluminal coronary intervention, or coronary artery bypass graft surgery within 12 weeks prior to Screening, or cerebrovascular accident within 24 weeks prior to Screening.
* Diabetes mellitus if newly diagnosed or if HbA1c ≥ 9.0%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of low density lipoprotein cholesterol (LDL-C). | 14 weeks
  Percent change in LDL-C from Baseline to week 14.

SECONDARY OUTCOMES:
Effect of ISIS 703802 on plasma angiopoietin like 3 (ANGPTL3). | 7 and 14 Weeks
  Absolute and percentage change in ANGPTL3 protein from Baseline to Week 14 will be summarized.
Effect of ISIS 703802 on lipid parameters. | 7 and 14 Weeks
  Absolute and percentage change from Baseline to Week 14 will be summarized.
Evaluate plasma trough levels of ISIS 703802. | 14 Weeks
  Plasma trough levels of ISIS 703802 during treatment period and those during post-treatment follow up period will be descriptively summarized.
The safety of ISIS 703802 by the incidence of treatment-emergent adverse events | 14 Weeks
  The safety of ISIS 703802 will be assessed by determining adverse effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Site, Québec, Quebec, Canada